CLINICAL TRIAL: NCT02795858
Title: A Phase II Study of Ramucirumab With Somatostatin Analog Therapy in Patients With Advanced, Progressive Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Jennifer Ang Chan, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-072
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Carcinoid Tumors
Keywords: Carcinoid Tumors
MeSH Terms: conditions — Carcinoid Tumor | interventions — Ramucirumab; Somatostatin; Octreotide; lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ramucirumab In Combination With Somatostatin Analog (Experimental): Patients will receive treatment with ramucirumab starting at a dose of 8 mg/kg intravenously every 14 days of a 28-day treatment cycle. Patients already receiving a somatostatin analog continued somatostatin analog therapy at their current dose. Patients not already receiving a somatostatin analog initiated treatment at an approved dose, according to institutional guidelines.
  Toxicity and adverse events will be examined in the first 10 patients who complete one cycle of therapy before expanding enrollment.
  Interventions: Drug: Ramucirumab; Drug: Somatostatin Analog

INTERVENTIONS:
Drug: Ramucirumab
  Other Names: Cyramza
Drug: Somatostatin Analog
  Other Names: octreotide; lanreotide

SUMMARY:
This research study is evaluating the drug Ramucirumab as a possible treatment for Advanced, Progressive Carcinoid Tumors.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. The purpose of this study is to test the safety and effectiveness of ramucirumab in advanced, progressive carcinoid tumors.

Cancer cells can make growth factors that cause the abnormal growth of new blood vessels. Ramucirumab is an investigational drug which works by blocking a receptor for a vascular growth factor, thereby preventing new blood vessels from forming. This may stop the cancer from growing or spreading and the tumor cells may die.

The FDA (the U.S. Food and Drug Administration) has not approved Ramucirumab for treatment of Carcinoid Tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed low- to intermediate-grade neuroendocrine tumor (carcinoid tumor).
* Carcinoid tumors of any site are eligible. Patients with pancreatic neuroendocrine tumors are excluded.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 10 for the evaluation of measurable disease.
* Locally advanced, unresectable or metastatic disease.
* Patients must have evidence of radiographic disease progression within the past 12 months. Progressive disease by RECIST criteria is not required.
* Age ≥ 18 years.
* ECOG performance status 0-1 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/ mm3
  * platelets ≥100,000/ mm3
  * hemoglobin ≥ 9 g/dL
  * total bilirubin ≤ 1.5 × institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional upper limit of normal, or ≤ 5× institutional upper limit of normal in the setting of liver metastases
  * creatinine ≤ 1.5 × upper limit of normal
  * urinary protein ≤ 1+ on dipstick or routine urinalysis (if urine dipstick or routine urinalysis is 2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours)
  * coagulation function Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) < 1.5 x institutional upper limit of normal. Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin.
  * The effects of ramucirumab on the developing human fetus are unknown. For this reason and because anti-antiangiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Ramucirumab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who have undergone major surgery within 28 days or subcutaneous venous access device placement within 7 days prior to study enrollment.
* Patients with elective or planned major surgery to be performed during the course of the clinical trial.
* Patients who are receiving any other investigational agents.
* Patients with any Grade 3-4 gastrointestinal bleeding within 3 months prior to enrollment.
* Patients with a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to registration.
* Patients who have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment.
* Patients with uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
* Patients who have congestive heart failure (NYHA Class III or IV), sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block within the six months preceding enrollment.
* Patients who have cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
* Patients with a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Patients receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Patients with uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
* Patients with symptomatic cholelithiasis.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Severely impaired lung function
  * Any active (acute or chronic) or uncontrolled infection/ disorders.
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
  * Psychiatric illness/social situations that would limit compliance with study requirement
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ramucirumab .
* Pregnant and breastfeeding women are excluded from this study because ramucirumab is associated with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ramucirumab, breastfeeding should be discontinued if the mother is treated with ramucirumab. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Chan, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez K, Kulke MH, Zheng H, Allen J, Clark J, Enzinger AC, Enzinger PC, Johnson BE, McCleary NJ, Parikh A, Patel A, Rubinson D, Yurgelun MB, Ramsey K, Johnson E, Graham C, Chan JA. A phase II study of ramucirumab and somatostatin analog therapy in patients with advanced neuroendocrine tumors. Oncologist. 2025 Jan 17;30(1):oyae364. doi: 10.1093/oncolo/oyae364. PMID 39834129

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab In Combination With Somatostatin Analog: Patients will receive treatment with Ramucirumab at a dose of 8mg/kg intravenously every 14 days of a 28-day treatment cycle.
  Patients will receive treatment with a Somatostatin Analog at a pre-determined dose.
Period: Overall Study
Arm/Group | Ramucirumab In Combination With Somatostatin Analog
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ramucirumab In Combination With Somatostatin Analog: Patients will receive treatment with Ramucirumab at a pre-determined dose intravenously every 14 days of a 28-day treatment cycle.
  Patients will receive treatment with a Somatostatin Analog at a pre-determined dose.
Arm/Group | Ramucirumab In Combination With Somatostatin Analog
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43
Primary Tumor Location [Count of Participants; unit: Participants]
  Small Intestine | 20
  Lung | 10
  Thymus | 3
  Rectum | 1
  Kidney | 1
  Unknown | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: To assess the progression-free survival duration of patients with advanced, progressive carcinoid tumors treated with ramucirumab in combination with somatostatin analog therapy. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Survival collected every 12 weeks in long-term follow-up. The median survival follow-up time was 23.5 months (range 1.7 - 76.6 months)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ramucirumab + Somatostatin Analog: Patients started treatment with ramucirumab at a dose of 8 mg/kg intravenously every 14 days of a 28-day treatment cycle. Patients already receiving a somatostatin analog continued somatostatin analog therapy at their current dose. Patients not already receiving a somatostatin analog initiated treatment at an approved dose, according to institutional guidelines.
Arm/Group | Ramucirumab + Somatostatin Analog
Number analyzed (Participants) | 43
months | 14.2 [9.0 to 25.6]

2. Secondary Outcome: Overall Survival
Description: To assess the overall survival duration of patients with advanced carcinoid tumors treated with ramucirumab. We will use the Kaplan-Meier method to estimate the distribution of overall survival.
Time Frame: The median survival follow-up time was 23.5 months (range 1.7 - 76.6 months)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ramucirumab + Somatostatin Analog: Patients will receive treatment with Ramucirumab starting at a dose of 8mg/kg intravenously every 14 days of a 28-day treatment cycle.
  Patients will receive treatment with a Somatostatin Analog at a pre-determined dose.
Arm/Group | Ramucirumab + Somatostatin Analog
Number analyzed (Participants) | 43
months | 24.9 [20.7 to 43.1]

3. Secondary Outcome: Overall Radiographic Response
Description: To evaluate disease response using RECIST criteria, version 1.1, of patients with advanced carcinoid tumors treated with Ramucirumab.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT include the following categories of disease response: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable disease (SD), less than 30% decrease but no more than 20% increase in sum of the longest diameter of target lesions.
  We will estimate the response rate and provide the associated 95% confidence interval.
Time Frame: 2 years
Population: Radiographic response rate was evaluated for all 43 eligible participants who started protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Somatostatin Analog
Number analyzed (Participants) | 43
Participants
  Partial Response | 2
  Stable Disease | 33
  Progressive Disease | 3
  Not Restaged | 5

4. Secondary Outcome: Biochemical Response (Chromogranin A)
Description: To evaluate biochemical response in patients with elevated chromogranin A at baseline, using levels of chromogranin-A measured at baseline and following treatment with Ramucirumab. Biochemical response was defined as greater than 50% drop in chromogranin A from baseline.
  During the screening period, all patients were evaluated for serum chromogranin A. Per protocol, if results of these are normal at baseline, they were not repeated while on study. If above institutional ULN at baseline, they were evaluated at time of tumor restaging.
Time Frame: 2 years
Population: 37 patients had an elevated chromogranin A level at baseline and were followed for biochemical response, as defined by a greater than 50% drop in chromogranin A level from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Somatostatin Analog
Number analyzed (Participants) | 37
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events evaluated on treatment on day 1 and 15 of each cycle and follow-up for 30 days off treatment. Observation period with median of 194 days and range (30-1416 days). All-Cause Mortality monitored/assessed up to 76.6 months
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Groups:
- Ramucirumab In Combination With Somatostatin Analog: Patients started treatment with ramucirumab at a dose of 8 mg/kg intravenously every 14 days of a 28-day treatment cycle. Patients already receiving a somatostatin analog continued somatostatin analog therapy at their current dose. Patients not already receiving a somatostatin analog initiated treatment at an approved dose, according to institutional guidelines.
Arm/Group | Ramucirumab In Combination With Somatostatin Analog
All-Cause Mortality (participants affected / at risk) | 33/43
Serious Adverse Events (participants affected / at risk) | 15/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramucirumab In Combination With Somatostatin Analog (N=43)
Pneumonia (Infections and infestations) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Cardiac chest pain (Cardiac disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
Intraventricular conduction (Cardiac disorders) | 1
Lower extremity edema (General disorders) | 1
Obstipation (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Pharyngeal dysphagia (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Small bowel obstruction (General disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab In Combination With Somatostatin Analog (N=43)
Abdominal pain (Gastrointestinal disorders) | 20
Alanine aminotransferase increased (Investigations) | 12
Alkaline phosphatase increased (Investigations) | 18
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 12
Aspartate aminotransferase increased (Investigations) | 26
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bloating (Gastrointestinal disorders) | 3
Blood bilirubin increased (Investigations) | 5
Bruising (Injury, poisoning and procedural complications) | 3
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Creatinine increased (Investigations) | 14
Dehydration (Metabolism and nutrition disorders) | 10
Diarrhea (Gastrointestinal disorders) | 23
Dizziness (Nervous system disorders) | 10
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Edema limbs (General disorders) | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 36
Flushing (Vascular disorders) | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 18
Hematuria (Renal and urinary disorders) | 10
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypertension (Vascular disorders) | 36
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypothyroidism (Endocrine disorders) | 4
Insomnia (Psychiatric disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Nausea (Gastrointestinal disorders) | 17
Neutrophil count decreased (Investigations) | 8
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 3 (6)
Platelet count decreased (Investigations) | 20
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Proteinuria (Renal and urinary disorders) | 26
Sinusitis (Infections and infestations) | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Tremor (Nervous system disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 9
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 9
Lower extremity swelling (General disorders) | 4
Abdominal cramping (Gastrointestinal disorders) | 3
Gum bleeding (General disorders) | 4
Early satiety (Gastrointestinal disorders) | 3
Hip pain (Musculoskeletal and connective tissue disorders) | 4
Hemoglobin decreased (Investigations) | 5
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT02795858/Prot_SAP_000.pdf